CLINICAL TRIAL: NCT00726388
Title: An Open-Label, Multiple-Dose, Multiple-Day, Non-Randomized, Single-Arm Safety Study Of Repeat-Doses Of DIC075V (Intravenous Diclofenac Sodium) In Patients With Acute Post-Operative Pain
Brief Title: An Open-Label Safety Study Of DIC075V (Intravenous Diclofenac Sodium) In Patients With Acute Post-Operative Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DFC-010; C1211011 (Other: Alias Study Number)
Record Dates: First submitted 2008-07-29; First posted 2008-07-31 (Estimated); Results first posted 2021-10-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-09

CONDITIONS: Pain, Postoperative
Keywords: safety; diclofenac; pain, postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- A (Experimental): IV administration of multiple doses of DIC075V (intravenous diclofenac sodium) over multiple days
  Interventions: Drug: DIC075V (intravenous diclofenac sodium)

INTERVENTIONS:
Drug: DIC075V (intravenous diclofenac sodium) — multiple doses up to 5 days

SUMMARY:
This is an open-label, multiple-dose, safety study of DIC075V in patients with acute post-operative pain following abdominal or orthopedic surgery.

DETAILED DESCRIPTION:
This is an open-label, multiple-dose, multiple-day, single-arm safety study of repeat-doses of DIC075V in patients with acute post-operative pain following abdominal (i.e., non-laparoscopic abdominal surgeries) or orthopedic (e.g., hip or knee joint replacement) surgery. Eligible patients will receive DIC075V IV bolus q6 hours. Safety assessments will be collected at baseline (immediately prior to starting DIC075V therapy) and at study discharge or early termination.

ELIGIBILITY:
Inclusion Criteria:

* abdominal ( non-laparoscopic abdominal surgeries) or orthopedic ( hip or knee joint replacement) surgery or other surgeries requiring multiple doses of parenterally administered NSAIDs over multiple days
* Expected stay > 48 hrs

Exclusion Criteria:

* bilirubin > 2.5 mg/dl
* prothrombin time is > 20% above the upper limit of normal
* serum creatinine is > 1.9 mg/dl at screening.
* known allergy or hypersensitivity to diclofenac, other NSAIDs,

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050 (Actual)
Dates: Start 2008-09-15 (Actual); Primary Completion 2009-05-08 (Actual); Study Completion 2009-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (45):
- United States (45):
  - West Alabama Research, LLC, Birmingham, Alabama
  - Alabama Clinical Therapeutics, Birmingham, Alabama
  - Shoals Clinical Research Associates, LLC, Eliza Coffee Memorial Hospital, Florence, Alabama
  - Horizon Research Group, Mobile, Alabama
  - Drug Research and Analysis Corp., Montgomery, Alabama
  - Jackson Hospital, Montgomery, Alabama
  - Helen Keller Memorial Hospital, Sheffield, Alabama
  - Pivotal Clinical Research, Peoria, Arizona
  - Precision Trials, Phoenix, Arizona
  - Teton Research, LLC, Little Rock, Arkansas
  - Vertex, Bakersfield, California
  - Lotus Clinical Research, Glendale, California
  - Physicians Clinical Research, Laguna Hills, California
  - National Institute of Clinical Research, Los Angeles, California
  - Lotus Clinical Research, Pasadena, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - North Coast Women's Care, Vista, California
  - American Clinical Research, Aurora, Colorado
  - Colorado Orthopedic Consultants, Englewood, Colorado
  - American Clinical Research Services, Steamboat Springs, Colorado
  - Orthopedic Associates of Hartford, Hartford, Connecticut
  - Nature Coast Clinical Research, Inverness, Florida
  - Sunrise Medical Research, Inc., Lauderdale Lakes, Florida
  - Pensacola Research Consultants, Pensacola, Florida
  - Florida Orthopedic Institute, Tampa, Florida
  - Soapstone Center for Clinical Research, Decatur, Georgia
  - JRSI Foundation The center for Hip and Knee Surgery, Mooresville, Indiana
  - University of Kansas Medical Center Department of Anesthesiology, Kansas City, Kansas
  - Validity Research, Merriam, Kansas
  - Tulane Univ. Medical Center, New Orleans, Louisiana
  - Great Falls Clinic, LLP, Great Falls, Montana
  - Albany Medical Center, Albany, New York
  - Staten Island University Hospital, Staten Island, New York
  - The Ohio State University Medical Center, Columbus, Ohio
  - Allegheny Pain Management, Altoona, Pennsylvania
  - University of Orthopedics Center, Altoona, Pennsylvania
  - Ilumina Clinical Associates, Johnstown, Pennsylvania
  - UPMC Presbyterian-Shadyshide Hospital, Pittsburgh, Pennsylvania
  - UPMC-St. Margaret's Hospital, Pittsburgh, Pennsylvania
  - Somerset Hospital, Somerset, Pennsylvania
  - University Orthopedics Center, State College, Pennsylvania
  - Comprehensive Pain Specialists, PLLC, Hendersonville, Tennessee
  - Endeavor Clinical Trials, San Antonio, Texas
  - Interventional Pain Management, San Antonio, Texas
  - Scott & White Clinic / Texas A&M Health Science Center, Temple, Texas

REFERENCES:
- [Derived] Chelly JE, Lacouture PG, Reyes CRD. Safety of Injectable HPbetaCD-Diclofenac in Older Patients with Acute Moderate-to-Severe Postoperative Pain: A Pooled Analysis of Three Phase III Trials. Drugs Aging. 2018 Mar;35(3):249-259. doi: 10.1007/s40266-018-0529-3. PMID 29492863

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with immediate acute postoperative pain, who were stable according to the study site's usual practice, were enrolled in the study. They received intravenous (IV) diclofenac sodium (DIC075V) bolus as their primary postoperative analgesic.
Pre-assignment Details: Total 1171 participants signed the inform consent form (ICF). Out of which 121 participants were screen failure and 1050 actually enrolled into the study and 971 assigned to study treatment.
Groups:
- DIC075V: Participants weighing greater than or equal to (>=) 95 kg received DIC075V 50 milligram (mg) IV bolus once every 6 hours. Participants with more than 1 non-steroidal anti-inflammatory drug (NSAIDS) related risk factor, example, weighing <95 kg along with mild renal insufficiency received DIC075V 37.5 mg IV bolus once every 6 hours. Participants received DIC075V for a minimum of 8 consecutive doses and until they were completely transitioned to oral analgesics, discharged from the institution, received a maximum of 5 days of treatment with DIC075V, or discontinued from the study, whichever occurred first. Participants returned to the clinic for a safety follow-up visit 4-10 days after their last dose of DIC075V and completed a safety follow-up telephone call 30-37 days post-last dose of DIC075V.
Period: Overall Study
Arm/Group | DIC075V
Started | 1050
Treated | 971
Completed | 943
Not Completed | 107
Not completed — Withdrawal by Subject | 5
Not completed — Adverse Event | 3
Not completed — Lost to Follow-up | 10
Not completed — Participants Non-compliant With Study Procedures | 5
Not completed — Other | 5
Not completed — Enrolled, Not Treated | 79

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received DIC075V and had at least 1 safety assessment.
Groups:
- DIC075V: Participants weighing >=95 kg received DIC075V 50 mg IV bolus once every 6 hours. Participants with more than 1 NSAIDS related risk factor, example, weighing <95 kg along with mild renal insufficiency received DIC075V 37.5 mg IV bolus once every 6 hours. Participants received DIC075V for a minimum of 8 consecutive doses and until they were completely transitioned to oral analgesics, discharged from the institution, received a maximum of 5 days of treatment with DIC075V, or discontinued from the study, whichever occurred first. Participants returned to the clinic for a safety follow-up visit 4-10 days after their last dose of DIC075V and completed a safety follow-up telephone call 30-37 days post-last dose of DIC075V.
Arm/Group | DIC075V
Number analyzed (Participants) | 971
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 617
  Male | 354

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. TEAEs were events between first dose of study drug and up to 37 days after last dose that were absent before treatment or that worsened relative to pretreatment state. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. TEAEs included SAEs and all non-SAEs that occurred during the study.
Time Frame: Day 1 of dosing up to maximum of 37 days after last dose (maximum up to 42 days)
Population: Safety population included all participants who received DIC075V and had at least 1 safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | DIC075V
Number analyzed (Participants) | 971
Participants
  TEAEs | 823
  SAEs | 73

2. Primary Outcome: Number of Participants Who Took at Least 1 Concomitant Medication
Description: Concomitant medications were medications that were taken concurrently on or after first dose of study drug.
Time Frame: Day 1 of dosing up to maximum of 37 days after last dose (maximum up to 42 days)
Population: Safety population included all participants who received DIC075V and had at least 1 safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | DIC075V
Number analyzed (Participants) | 971
Participants | 971

3. Primary Outcome: Number of Participants With Abnormal Urinalysis Findings
Description: Urine parameters included gravity, glucose, protein, and bilirubin. Abnormalities were judged by the investigator.
Time Frame: Baseline (Day 1, immediately before dosing) up to study discharge/early termination (maximum up to Day 5)
Population: Safety population included all participants who received DIC075V and had at least 1 safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | DIC075V
Number analyzed (Participants) | 971
Participants | 2

4. Primary Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Abnormalities at Baseline
Description: 12-lead ECG parameters were evaluated. Clinically significant abnormal ECG findings were based on investigator's discretion.
Time Frame: Baseline (Day 1, immediately before dosing)
Population: Safety population included all participants who received DIC075V and had at least 1 safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | DIC075V
Number analyzed (Participants) | 971
Participants | 14

5. Primary Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Abnormalities at Study Discharge/Early Termination
Description: as for outcome 4
Time Frame: Study discharge/early termination (maximum up to Day 5)
Population: Safety population included all participants who received DIC075V and had at least 1 safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | DIC075V
Number analyzed (Participants) | 971
Participants | 13

6. Primary Outcome: Change From Baseline in Blood Pressure at Study Discharge/Early Termination
Description: Change from baseline in systolic blood pressure (SBP) and diastolic blood pressure (DBP) in millimeter of mercury (mmHg) was reported. The blood pressure was assessed after the participant had taken rest for 5 minutes.
Time Frame: Baseline (Day 1, immediately before dosing), Study discharge/early termination (maximum up to 5 days)
Population: Safety population included all participants who received DIC075V and had at least 1 safety assessment. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | DIC075V
Number analyzed (Participants) | 958
mmHg
  SBP | -2.2 (21.5)
  DBP | -0.5 (14.7)

7. Primary Outcome: Change From Baseline in Blood Pressure at Clinic Follow-up Visit
Description: Change from baseline in SBP and DBP in mmHg was reported. The blood pressure was assessed after the participant had taken rest for 5 minutes.
Time Frame: Baseline (Day 1, immediately before dosing), Clinic follow-up visit (4-10 days after last dose, maximum up to 15 days)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | DIC075V
Number analyzed (Participants) | 941
mmHg
  SBP | 0.2 (21.4)
  DBP | 4.4 (13.9)

8. Primary Outcome: Change From Baseline in Respiratory Rate at Study Discharge/Early Termination
Description: Respiratory rate was measured after the participant had taken rest for 5 minutes.
Time Frame: Baseline (Day 1, immediately before dosing), Study discharge/early termination (maximum up to 5 days)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | DIC075V
Number analyzed (Participants) | 957
Breaths per minute | 1.3 (3.0)

9. Primary Outcome: Change From Baseline in Respiratory Rate at Clinic Follow-up Visit
Description: Respiratory rate was measured after the participant had taken rest for 5 minutes.
Time Frame: Baseline (Day 1, immediately before dosing), Clinic follow-up visit (4-10 days after last dose, maximum up to 15 days)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | DIC075V
Number analyzed (Participants) | 937
Breaths per minute | 1.0 (3.8)

10. Primary Outcome: Change From Baseline in Heart Rate at Study Discharge/Early Termination
Description: Change from baseline in heart rate in beats per minute was reported. The heart rate was assessed after the participant had taken rest for 5 minutes.
Time Frame: Baseline (Day 1, immediately before dosing), Study discharge/early termination (maximum up to 5 days)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | DIC075V
Number analyzed (Participants) | 958
Beats per minute | 3.8 (15.4)

11. Primary Outcome: Change From Baseline in Heart Rate at Clinic Follow-up Visit
Description: as for outcome 10
Time Frame: Baseline (Day 1, immediately before dosing), Clinic follow-up visit (4-10 days after last dose, maximum up to 15 days)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | DIC075V
Number analyzed (Participants) | 939
Beats per minute | 2.4 (15.5)

12. Primary Outcome: Number of Participants With Wound Assessment at Study Discharge/Early Termination
Description: Wound assessment had 6 questions, completed by investigator/sub-investigator. Question related to extent of healing; extent and degree of inflammation and extent of drainage had options: much better than expected, better than expected, normal, slower than expected, and much slower than expected. Question related to separation of surgical incision had options: no separation, barely detectible separation, localized separation, mostly separated, and complete separation (dehiscence). Question related to infection at surgical site had options: definitely, no infection, possibly infected, probably infected, certainly infected, and abscess/gross cellulitis. Question related to prescription of postoperative systemic antibiotics had options: no, yes for prophylaxis, and yes for infection. Every question there was category "Not Done" for participants with no wound assessment other than the reason 'missing' and category "Missing", where participants were missing for wound assessment.
Time Frame: Study discharge/early termination (maximum up to Day 5)
Population: Safety population included all participants who received DIC075V and had at least 1 safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | DIC075V
Number analyzed (Participants) | 971
Participants
  Extent of healing: Much better than expected | 40
  Extent of healing: Better than expected | 154
  Extent of healing: Normal | 727
  Extent of healing: Slower than expected | 11
  Extent of healing: Much slower than expected | 0
  Extent of healing: Not done | 33
  Extent of healing: Missing | 6
  Extent and degree of Inflammation: Much better than expected | 50
  Extent and degree of inflammation: Better than expected | 214
  Extent and degree of Inflammation: Normal | 657
  Extent and degree of Inflammation: Slower than expected | 11
  Extent and degree of Inflammation: Much slower than expected | 0
  Extent and degree of inflammation: Not done | 33
  Extent and degree of inflammation: Missing | 6
  Extent of drainage: Much better than expected | 78
  Extent of drainage: Better than expected | 195
  Extent of drainage: Normal | 633
  Extent of drainage: Slower than expected | 29
  Extent of drainage: Much slower than expected | 1
  Extent of drainage: Not done | 33
  Extent of drainage: Missing | 2
  Separation of Incision: No separation | 809
  Separation of Incision: Barely detectable separation | 87
  Separation of incision: Localized separation | 35
  Separation of incision: Mostly separated | 0
  Separation of incision: Complete separation | 0
  Separation of incision: Not done | 33
  Separation of incision: Missing | 7
  Infection at surgical site: Definitely, No infection | 921
  Infection at surgical site: Possibly infected | 12
  Infection at surgical site: Probably infected | 1
  Infection at surgical site: Certainly infected | 1
  Infection at surgical site: Abscess or gross cellulitis | 0
  Infection at surgical site: Not done | 33
  Infection at surgical site: Missing | 3
  Postoperative systemic antibiotics: No | 673
  Postoperative systemic antibiotics: Yes, for prophylaxis | 262
  Postoperative systemic antibiotics: Yes, for infection | 1
  Postoperative systemic antibiotics: Not done | 33
  Postoperative systemic antibiotics: Missing | 2

13. Primary Outcome: Number of Participants With Thrombophlebitis Assessment Evaluation at Baseline
Description: Thrombophlebitis assessment evaluation was done using following grades: 0 equals to (=) no reaction, 1= tenderness along the vein, 2= continuous tenderness of pain with redness, 3= palpable swelling or thrombosis within length of cannula, 4= palpable swelling or thrombosis beyond the length of the cannula and 5= palpable swelling or thrombosis beyond the length of the cannula with overt infection.
Time Frame: Baseline (Day 1, immediately before dosing)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | DIC075V
Number analyzed (Participants) | 963
Participants
  Grade 0 | 960
  Grade 1 | 3
  Grade 2 | 0
  Grade 3 | 0
  Grade 4 | 0
  Grade 5 | 0

14. Primary Outcome: Number of Participants With Thrombophlebitis Assessment Evaluation at Study Discharge/Early Termination
Description: Thrombophlebitis assessment evaluation was done using following grades: 0= no reaction, 1= tenderness along the vein, 2= continuous tenderness of pain with redness, 3= palpable swelling or thrombosis within length of cannula, 4= palpable swelling or thrombosis beyond the length of the cannula and 5= palpable swelling or thrombosis beyond the length of the cannula with overt infection.
Time Frame: Study discharge/early termination (maximum up to Day 5)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | DIC075V
Number analyzed (Participants) | 957
Participants
  Grade 0 | 925
  Grade 1 | 26
  Grade 2 | 3
  Grade 3 | 3
  Grade 4 | 0
  Grade 5 | 0

15. Primary Outcome: Number of Participants With Clinically Significant Physical Examination Abnormalities at Screening
Description: Physical examination included the assessment of general appearance, skin; head, ears, eyes, nose, and throat (HEENT); neck/thyroid; oral cavity; lymph nodes; cardiovascular; lungs; abdomen; genitourinary; neurologic and joints/extremities. Clinically significant physical examination findings were based on investigator's discretion.
Time Frame: Screening (0 to 21 days prior to surgery)
Population: Safety population included all participants who had received DIC075V and had at least 1 safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | DIC075V
Number analyzed (Participants) | 971
Participants
  General Appearance | 8
  Skin | 3
  HEENT | 7
  Neck/Thyroid | 1
  Oral Cavity | 2
  Lymph Nodes | 0
  Cardiovascular | 3
  Lungs | 0
  Breasts | 0
  Abdomen | 29
  Genitourinary | 32
  Neurologic | 10
  Joints/Extremities | 295

16. Primary Outcome: Number of Participants With Clinically Significant Physical Examination Abnormalities at Clinic Follow-up Visit
Description: Physical examination included the assessment of general appearance, skin; HEENT; neck/thyroid; oral cavity; lymph nodes; cardiovascular; lungs; abdomen; genitourinary; neurologic and joints/extremities. Clinically significant physical examination findings were based on investigator's discretion.
Time Frame: Clinic follow-up visit (4-10 days after last dose, maximum up to 15 days)
Population: Safety population included all participants who had received DIC075V and had at least 1 safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | DIC075V
Number analyzed (Participants) | 971
Participants
  General appearance | 8
  Skin | 13
  HEENT | 2
  Neck/Thyroid | 1
  Oral Cavity | 0
  Lymph Nodes | 0
  Cardiovascular | 5
  Lungs | 5
  Breasts | 0
  Abdomen | 12
  Genitourinary | 1
  Neurologic | 5
  Joints/Extremities | 41

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study. Any clinical significant changes in laboratory examinations were reported as AEs. Safety population included all participants who had received DIC075V and had at least 1 safety assessment.
Arm/Group | DIC075V
Serious Adverse Events (participants affected / at risk) | 73/971
Other Adverse Events (participants affected / at risk) | 816/971
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DIC075V (N=971)
ATRIAL FIBRILLATION (Cardiac disorders) | 2
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 3
NAUSEA (Gastrointestinal disorders) | 2
VOMITING (Gastrointestinal disorders) | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 1
ANAL HAEMORRHAGE (Gastrointestinal disorders) | 1
CONSTIPATION (Gastrointestinal disorders) | 1
ENTEROCUTANEOUS FISTULA (Gastrointestinal disorders) | 1
HAEMATOCHEZIA (Gastrointestinal disorders) | 1
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1
PANCREATITIS (Gastrointestinal disorders) | 1
PERITONITIS (Gastrointestinal disorders) | 1
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1
PYREXIA (General disorders) | 2
NON-CARDIAC CHEST PAIN (General disorders) | 1
OEDEMA PERIPHERAL (General disorders) | 1
INCISION SITE CELLULITIS (Infections and infestations) | 3
WOUND INFECTION (Infections and infestations) | 3
CELLULITIS (Infections and infestations) | 2
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 2
SEPSIS (Infections and infestations) | 2
ABDOMINAL WALL ABSCESS (Infections and infestations) | 1
BRONCHITIS (Infections and infestations) | 1
CATHETER SEPSIS (Infections and infestations) | 1
HAEMATOMA INFECTION (Infections and infestations) | 1
INCISION SITE ABSCESS (Infections and infestations) | 1
INCISION SITE INFECTION (Infections and infestations) | 1
LOBAR PNEUMONIA (Infections and infestations) | 1
PELVIC ABSCESS (Infections and infestations) | 1
POST PROCEDURAL CELLULITIS (Infections and infestations) | 1
VAGINAL CELLULITIS (Infections and infestations) | 1
WOUND ABSCESS (Infections and infestations) | 1
WOUND INFECTION STAPHYLOCOCCAL (Infections and infestations) | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 5
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 2
ANASTOMOTIC HAEMORRHAGE (Injury, poisoning and procedural complications) | 1
ANASTOMOTIC LEAK (Injury, poisoning and procedural complications) | 1
CONTUSION (Injury, poisoning and procedural complications) | 1
INCISION SITE HAEMATOMA (Injury, poisoning and procedural complications) | 1
INCISION SITE PAIN (Injury, poisoning and procedural complications) | 1
POST PROCEDURAL DISCHARGE (Injury, poisoning and procedural complications) | 1
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1
POSTOPERATIVE ILEUS (Injury, poisoning and procedural complications) | 1
POSTOPERATIVE WOUND COMPLICATION (Injury, poisoning and procedural complications) | 1
TENDON RUPTURE (Injury, poisoning and procedural complications) | 1
BLOOD CREATININE INCREASED (Investigations) | 3
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 2
BLOOD CULTURE POSITIVE (Investigations) | 1
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 1
LIVER FUNCTION TEST ABNORMAL (Investigations) | 1
DEHYDRATION (Metabolism and nutrition disorders) | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 1
BENIGN SMALL INTESTINAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
SEDATION (Nervous system disorders) | 2
MENTAL STATUS CHANGES (Psychiatric disorders) | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 2
RENAL FAILURE (Renal and urinary disorders) | 1
RENAL TUBULAR NECROSIS (Renal and urinary disorders) | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 6
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 2
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 1
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 1
HYPOTENSION (Vascular disorders) | 1
BACTERAEMIA (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DIC075V (N=971)
ANAEMIA (Blood and lymphatic system disorders) | 8
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 11
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 11
HAEMORRHAGIC ANAEMIA (Blood and lymphatic system disorders) | 3
COAGULOPATHY (Blood and lymphatic system disorders) | 2
THROMBOCYTHAEMIA (Blood and lymphatic system disorders) | 1
BRADYCARDIA (Cardiac disorders) | 10
ATRIAL FIBRILLATION (Cardiac disorders) | 6
TACHYCARDIA (Cardiac disorders) | 32
SINUS TACHYCARDIA (Cardiac disorders) | 4
SINUS BRADYCARDIA (Cardiac disorders) | 3
ANGINA PECTORIS (Cardiac disorders) | 2
ARRHYTHMIA (Cardiac disorders) | 2
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1
CARDIOMEGALY (Cardiac disorders) | 2
MYOCARDIAL INFARCTION (Cardiac disorders) | 2
SUPRAVENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 2
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 1
BUNDLE BRANCH BLOCK LEFT (Cardiac disorders) | 1
BUNDLE BRANCH BLOCK RIGHT (Cardiac disorders) | 1
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1
PALPITATIONS (Cardiac disorders) | 1
PERICARDIAL EFFUSION (Cardiac disorders) | 1
RIGHT VENTRICULAR HYPERTROPHY (Cardiac disorders) | 1
TINNITUS (Ear and labyrinth disorders) | 1
GOITRE (Endocrine disorders) | 1
CONJUNCTIVITIS (Eye disorders) | 1
DRY EYE (Eye disorders) | 1
EYE IRRITATION (Eye disorders) | 1
EYE PAIN (Eye disorders) | 1
EYELID DISORDER (Eye disorders) | 1
VISION BLURRED (Eye disorders) | 1
NAUSEA (Gastrointestinal disorders) | 359
CONSTIPATION (Gastrointestinal disorders) | 181
VOMITING (Gastrointestinal disorders) | 81
FLATULENCE (Gastrointestinal disorders) | 38
DYSPEPSIA (Gastrointestinal disorders) | 36
DIARRHOEA (Gastrointestinal disorders) | 28
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 16
DRY MOUTH (Gastrointestinal disorders) | 11
ABDOMINAL PAIN (Gastrointestinal disorders) | 7
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 5
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 3
HAEMATOCHEZIA (Gastrointestinal disorders) | 2
STOMACH DISCOMFORT (Gastrointestinal disorders) | 3
GASTRITIS (Gastrointestinal disorders) | 2
HAEMORRHOIDS (Gastrointestinal disorders) | 2
LIP DRY (Gastrointestinal disorders) | 2
RETCHING (Gastrointestinal disorders) | 2
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1
ABDOMINAL TENDERNESS (Gastrointestinal disorders) | 1
ANAL ULCER (Gastrointestinal disorders) | 1
ASCITES (Gastrointestinal disorders) | 1
COLONIC POLYP (Gastrointestinal disorders) | 1
EPIGASTRIC DISCOMFORT (Gastrointestinal disorders) | 1
ERUCTATION (Gastrointestinal disorders) | 1
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 1
HAEMATEMESIS (Gastrointestinal disorders) | 1
ILEUS (Gastrointestinal disorders) | 1
ILEUS PARALYTIC (Gastrointestinal disorders) | 1
LIP ULCERATION (Gastrointestinal disorders) | 1
PARAESTHESIA ORAL (Gastrointestinal disorders) | 1
RECTAL DISCHARGE (Gastrointestinal disorders) | 1
SWOLLEN TONGUE (Gastrointestinal disorders) | 1
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1
TONGUE BLISTERING (Gastrointestinal disorders) | 1
TONGUE DISORDER (Gastrointestinal disorders) | 1
TOOTHACHE (Gastrointestinal disorders) | 1
PYREXIA (General disorders) | 56
INFUSION SITE PAIN (General disorders) | 50
OEDEMA PERIPHERAL (General disorders) | 37
ASTHENIA (General disorders) | 25
INFUSION SITE EXTRAVASATION (General disorders) | 14
CHILLS (General disorders) | 12
HYPOTHERMIA (General disorders) | 12
INFUSION SITE THROMBOSIS (General disorders) | 6
FATIGUE (General disorders) | 4
GENERALISED OEDEMA (General disorders) | 4
INFUSION SITE ERYTHEMA (General disorders) | 4
INFUSION SITE SWELLING (General disorders) | 4
BREAKTHROUGH PAIN (General disorders) | 3
CHEST PAIN (General disorders) | 3
INFUSION SITE OEDEMA (General disorders) | 3
CHEST DISCOMFORT (General disorders) | 2
INFUSION SITE IRRITATION (General disorders) | 2
OEDEMA (General disorders) | 2
ADVERSE DRUG REACTION (General disorders) | 1
APPLICATION SITE VESICLES (General disorders) | 1
EARLY SATIETY (General disorders) | 1
FACE OEDEMA (General disorders) | 1
FEELING HOT (General disorders) | 1
IMPAIRED HEALING (General disorders) | 1
INFUSION SITE BRUISING (General disorders) | 1
INFUSION SITE HAEMATOMA (General disorders) | 1
INFUSION SITE HAEMORRHAGE (General disorders) | 1
INFUSION SITE PARAESTHESIA (General disorders) | 1
INFUSION SITE WARMTH (General disorders) | 1
INJECTION SITE HAEMORRHAGE (General disorders) | 1
INJECTION SITE PAIN (General disorders) | 1
INJECTION SITE SWELLING (General disorders) | 1
PAIN (General disorders) | 1
PITTING OEDEMA (General disorders) | 1
THIRST (General disorders) | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 1
URINARY TRACT INFECTION (Infections and infestations) | 20
WOUND INFECTION (Infections and infestations) | 9
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 4
CELLULITIS (Infections and infestations) | 3
INCISION SITE INFECTION (Infections and infestations) | 4
NASOPHARYNGITIS (Infections and infestations) | 5
INCISION SITE ABSCESS (Infections and infestations) | 3
PNEUMONIA (Infections and infestations) | 4
SINUSITIS (Infections and infestations) | 4
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4
BRONCHITIS (Infections and infestations) | 2
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 3
BACTERAEMIA (Infections and infestations) | 1
CANDIDIASIS (Infections and infestations) | 2
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 2
FUNGAL INFECTION (Infections and infestations) | 2
GASTROENTERITIS VIRAL (Infections and infestations) | 2
WOUND INFECTION STAPHYLOCOCCAL (Infections and infestations) | 1
ANAL TINEA (Infections and infestations) | 1
CYSTITIS (Infections and infestations) | 1
FOLLICULITIS (Infections and infestations) | 1
GASTROENTERITIS (Infections and infestations) | 1
INFECTION (Infections and infestations) | 1
KIDNEY INFECTION (Infections and infestations) | 1
ORAL HERPES (Infections and infestations) | 1
OSTEOMYELITIS ACUTE (Infections and infestations) | 1
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1
TINEA PEDIS (Infections and infestations) | 1
TOOTH ABSCESS (Infections and infestations) | 1
ANAEMIA POSTOPERATIVE (Injury, poisoning and procedural complications) | 218
INCISION SITE COMPLICATION (Injury, poisoning and procedural complications) | 13
POST PROCEDURAL OEDEMA (Injury, poisoning and procedural complications) | 12
INCISION SITE ERYTHEMA (Injury, poisoning and procedural complications) | 9
POST PROCEDURAL DISCHARGE (Injury, poisoning and procedural complications) | 8
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 6
INCISION SITE HAEMORRHAGE (Injury, poisoning and procedural complications) | 7
CONTUSION (Injury, poisoning and procedural complications) | 5
FALL (Injury, poisoning and procedural complications) | 6
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 3
INCISION SITE OEDEMA (Injury, poisoning and procedural complications) | 3
PROCEDURAL HYPOTENSION (Injury, poisoning and procedural complications) | 3
SEROMA (Injury, poisoning and procedural complications) | 3
SKIN LACERATION (Injury, poisoning and procedural complications) | 3
EXCORIATION (Injury, poisoning and procedural complications) | 2
INCISION SITE PAIN (Injury, poisoning and procedural complications) | 1
POSTOPERATIVE WOUND COMPLICATION (Injury, poisoning and procedural complications) | 1
PROCEDURAL NAUSEA (Injury, poisoning and procedural complications) | 2
ESCHAR (Injury, poisoning and procedural complications) | 1
FRACTURE (Injury, poisoning and procedural complications) | 1
HIP FRACTURE (Injury, poisoning and procedural complications) | 1
INCISION SITE BLISTER (Injury, poisoning and procedural complications) | 1
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 1
LIGAMENT RUPTURE (Injury, poisoning and procedural complications) | 1
PROCEDURAL HYPERTENSION (Injury, poisoning and procedural complications) | 1
PROCEDURAL SITE REACTION (Injury, poisoning and procedural complications) | 1
PROCEDURAL VOMITING (Injury, poisoning and procedural complications) | 1
THERMAL BURN (Injury, poisoning and procedural complications) | 1
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 1
WOUND SECRETION (Injury, poisoning and procedural complications) | 1
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 61
PROTHROMBIN TIME PROLONGED (Investigations) | 14
BLOOD CREATININE INCREASED (Investigations) | 7
URINE OUTPUT DECREASED (Investigations) | 10
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 8
BREATH SOUNDS ABNORMAL (Investigations) | 8
OXYGEN SATURATION DECREASED (Investigations) | 7
BODY TEMPERATURE INCREASED (Investigations) | 6
LIVER FUNCTION TEST ABNORMAL (Investigations) | 5
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 5
BLOOD AMYLASE INCREASED (Investigations) | 5
BLOOD GLUCOSE INCREASED (Investigations) | 5
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 4
LIPASE INCREASED (Investigations) | 4
BLOOD BILIRUBIN INCREASED (Investigations) | 3
BLOOD MAGNESIUM DECREASED (Investigations) | 3
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 3
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 3
BLOOD CREATINE PHOSPHOKINASE MB INCREASED (Investigations) | 2
BLOOD UREA INCREASED (Investigations) | 2
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 1
HEART RATE IRREGULAR (Investigations) | 2
PLATELET COUNT DECREASED (Investigations) | 2
RESPIRATORY RATE DECREASED (Investigations) | 2
RESPIRATORY RATE INCREASED (Investigations) | 2
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 2
BLOOD ALBUMIN DECREASED (Investigations) | 2
BLOOD ALBUMIN INCREASED (Investigations) | 1
BLOOD ALKALINE PHOSPHATASE (Investigations) | 1
BLOOD ALKALINE PHOSPHATASE DECREASED (Investigations) | 1
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 1
BLOOD PRESSURE DECREASED (Investigations) | 1
BLOOD PRESSURE INCREASED (Investigations) | 1
BLOOD URINE PRESENT (Investigations) | 1
CAROTID BRUIT (Investigations) | 1
CHEST X-RAY ABNORMAL (Investigations) | 1
CREATININE RENAL CLEARANCE DECREASED (Investigations) | 1
ELECTROCARDIOGRAM ST SEGMENT ABNORMAL (Investigations) | 1
ELECTROCARDIOGRAM T WAVE ABNORMAL (Investigations) | 1
FIBRIN D DIMER INCREASED (Investigations) | 1
HAEMATOCRIT DECREASED (Investigations) | 1
HAEMOGLOBIN DECREASED (Investigations) | 1
HEART RATE INCREASED (Investigations) | 1
HEPATIC ENZYME INCREASED (Investigations) | 1
PROTEIN TOTAL DECREASED (Investigations) | 1
PROTEIN TOTAL INCREASED (Investigations) | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 37
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 13
HYPONATRAEMIA (Metabolism and nutrition disorders) | 13
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 9
HYPERKALAEMIA (Metabolism and nutrition disorders) | 5
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 5
DEHYDRATION (Metabolism and nutrition disorders) | 3
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 4
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 4
HYPOPROTEINAEMIA (Metabolism and nutrition disorders) | 4
ANOREXIA (Metabolism and nutrition disorders) | 3
DECREASED APPETITE (Metabolism and nutrition disorders) | 3
DIABETES MELLITUS (Metabolism and nutrition disorders) | 3
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 2
HYPOCHLORAEMIA (Metabolism and nutrition disorders) | 2
FLUID RETENTION (Metabolism and nutrition disorders) | 1
GOUT (Metabolism and nutrition disorders) | 1
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 1
HYPERMAGNESAEMIA (Metabolism and nutrition disorders) | 1
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 1
IMPAIRED FASTING GLUCOSE (Metabolism and nutrition disorders) | 1
KWASHIORKOR (Metabolism and nutrition disorders) | 1
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 1
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 1
VITAMIN B12 DEFICIENCY (Metabolism and nutrition disorders) | 1
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 34
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 16
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 6
BACK PAIN (Musculoskeletal and connective tissue disorders) | 7
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 7
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 6
MUSCLE TIGHTNESS (Musculoskeletal and connective tissue disorders) | 3
NECK PAIN (Musculoskeletal and connective tissue disorders) | 3
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 2
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 2
ARTHROFIBROSIS (Musculoskeletal and connective tissue disorders) | 1
COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 1
EXOSTOSIS (Musculoskeletal and connective tissue disorders) | 1
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 1
HYPERCREATINAEMIA (Musculoskeletal and connective tissue disorders) | 1
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 1
JOINT RANGE OF MOTION DECREASED (Musculoskeletal and connective tissue disorders) | 1
LIMB DISCOMFORT (Musculoskeletal and connective tissue disorders) | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 1
NECK MASS (Musculoskeletal and connective tissue disorders) | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
THYROID NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
HEADACHE (Nervous system disorders) | 56
DIZZINESS (Nervous system disorders) | 49
HYPOAESTHESIA (Nervous system disorders) | 12
SOMNOLENCE (Nervous system disorders) | 8
PARAESTHESIA (Nervous system disorders) | 6
PERONEAL NERVE PALSY (Nervous system disorders) | 4
LETHARGY (Nervous system disorders) | 3
SEDATION (Nervous system disorders) | 1
NEUROPATHY PERIPHERAL (Nervous system disorders) | 2
SINUS HEADACHE (Nervous system disorders) | 2
SYNCOPE (Nervous system disorders) | 2
AURA (Nervous system disorders) | 1
CAROTID ARTERY STENOSIS (Nervous system disorders) | 1
DYSGEUSIA (Nervous system disorders) | 1
ENCEPHALOPATHY (Nervous system disorders) | 1
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1
MEMORY IMPAIRMENT (Nervous system disorders) | 1
MOTOR DYSFUNCTION (Nervous system disorders) | 1
NERVE COMPRESSION (Nervous system disorders) | 1
SYNCOPE VASOVAGAL (Nervous system disorders) | 1
TREMOR (Nervous system disorders) | 1
INSOMNIA (Psychiatric disorders) | 130
ANXIETY (Psychiatric disorders) | 22
CONFUSIONAL STATE (Psychiatric disorders) | 9
MENTAL STATUS CHANGES (Psychiatric disorders) | 3
AGITATION (Psychiatric disorders) | 3
DEPRESSION (Psychiatric disorders) | 3
HALLUCINATION (Psychiatric disorders) | 3
RESTLESSNESS (Psychiatric disorders) | 3
ABNORMAL DREAMS (Psychiatric disorders) | 1
DELIRIUM TREMENS (Psychiatric disorders) | 1
DISORIENTATION (Psychiatric disorders) | 1
FLAT AFFECT (Psychiatric disorders) | 1
HALLUCINATION, VISUAL (Psychiatric disorders) | 1
NIGHTMARE (Psychiatric disorders) | 1
URINARY RETENTION (Renal and urinary disorders) | 21
RENAL FAILURE ACUTE (Renal and urinary disorders) | 5
BLADDER SPASM (Renal and urinary disorders) | 6
DYSURIA (Renal and urinary disorders) | 4
HAEMATURIA (Renal and urinary disorders) | 3
RENAL FAILURE (Renal and urinary disorders) | 2
INCONTINENCE (Renal and urinary disorders) | 2
OLIGURIA (Renal and urinary disorders) | 2
URINARY INCONTINENCE (Renal and urinary disorders) | 2
ANURIA (Renal and urinary disorders) | 1
AZOTAEMIA (Renal and urinary disorders) | 1
BLADDER DISCOMFORT (Renal and urinary disorders) | 1
BLADDER DISORDER (Renal and urinary disorders) | 1
RENAL CYST (Renal and urinary disorders) | 1
RENAL DISORDER (Renal and urinary disorders) | 1
UROGENITAL FISTULA (Renal and urinary disorders) | 1
TESTICULAR OEDEMA (Reproductive system and breast disorders) | 1
VAGINAL DISCHARGE (Reproductive system and breast disorders) | 1
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 1
VULVOVAGINAL BURNING SENSATION (Reproductive system and breast disorders) | 1
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 28
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 15
COUGH (Respiratory, thoracic and mediastinal disorders) | 14
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 11
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 4
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 6
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 5
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 6
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 4
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 3
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 3
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 3
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 2
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2
NASAL DRYNESS (Respiratory, thoracic and mediastinal disorders) | 2
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY DEPRESSION (Respiratory, thoracic and mediastinal disorders) | 2
TACHYPNOEA (Respiratory, thoracic and mediastinal disorders) | 2
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 1
NASAL DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 1
PHARYNGEAL OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 1
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY GRANULOMA (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1
RALES (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 1
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1
SPUTUM DISCOLOURED (Respiratory, thoracic and mediastinal disorders) | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 125
BLISTER (Skin and subcutaneous tissue disorders) | 11
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 9
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 7
RASH (Skin and subcutaneous tissue disorders) | 7
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 6
ERYTHEMA (Skin and subcutaneous tissue disorders) | 4
DERMATITIS (Skin and subcutaneous tissue disorders) | 3
SKIN DISCOLOURATION (Skin and subcutaneous tissue disorders) | 2
ALOPECIA (Skin and subcutaneous tissue disorders) | 1
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 1
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 1
DRY SKIN (Skin and subcutaneous tissue disorders) | 1
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 1
ECZEMA (Skin and subcutaneous tissue disorders) | 1
HYPOAESTHESIA FACIAL (Skin and subcutaneous tissue disorders) | 1
INGROWING NAIL (Skin and subcutaneous tissue disorders) | 1
LEUKOCYTOCLASTIC VASCULITIS (Skin and subcutaneous tissue disorders) | 1
PSORIASIS (Skin and subcutaneous tissue disorders) | 1
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 1
ROSACEA (Skin and subcutaneous tissue disorders) | 1
STASIS DERMATITIS (Skin and subcutaneous tissue disorders) | 1
SWELLING FACE (Skin and subcutaneous tissue disorders) | 1
URTICARIA (Skin and subcutaneous tissue disorders) | 1
HYPOTENSION (Vascular disorders) | 59
HYPERTENSION (Vascular disorders) | 33
DEEP VEIN THROMBOSIS (Vascular disorders) | 3
FLUSHING (Vascular disorders) | 3
WOUND HAEMORRHAGE (Vascular disorders) | 3
DIASTOLIC HYPOTENSION (Vascular disorders) | 2
HAEMATOMA (Vascular disorders) | 2
HOT FLUSH (Vascular disorders) | 2
HYPERTENSIVE CRISIS (Vascular disorders) | 1
PALLOR (Vascular disorders) | 1
VAGINAL INFECTION (Infections and infestations) | 1
INCISION SITE HAEMATOMA (Injury, poisoning and procedural complications) | 1
DEPRESSION POSTOPERATIVE (Injury, poisoning and procedural complications) | 1
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 1
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.